CLINICAL TRIAL: NCT02985827
Title: An Open-Label, Single-Center Study to Evaluate Symptom Response and Tear Film Cooling Dynamics of Normal and Dry Eye Patients Secondary to Application of a Menthol-Containing Eyedrop (Rohto® Hydra)
Brief Title: Symptom Response in Normal and Dry Eye Patients Secondary to Application of a Menthol-Containing Eyedrop (Rohto® Hydra)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Menthol FLIR
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2016-12

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rohto (r) Hydra (Active Comparator): Menthol containing over the counter eyedrop
  Interventions: Drug: Rohto (r) Hydra; Drug: Systane (r) Ultra
- Systane (r) Ultra (Placebo Comparator): Non-Menthol containing over the counter eyedrop
  Interventions: Drug: Rohto (r) Hydra; Drug: Systane (r) Ultra

INTERVENTIONS:
Drug: Rohto (r) Hydra — Rohto (r) Hydra; Over the counter Eyedrop, 1 gtt OU single-masked in-office dose
  Other Names: Rohto Hydra
Drug: Systane (r) Ultra — Systane (r) Ultra; Over the counter Eyedrop, 1 gtt OU single-masked in-office dose
  Other Names: Systane Ultra

SUMMARY:
The purpose of the study is to analyze the sensation to eye drops containing menthol in people with healthy eyes and in people with dry eyes. This study also examines the temperature of your eye using an Infrared Camera.

DETAILED DESCRIPTION:
Dry eye disease (DED) has been defined as a multifactorial disease of the tears and ocular surface that results in symptoms of discomfort, visual disturbance, and tear film instability with potential damage to the ocular surface. It is accompanied by increased osmolarity of the tear film and inflammation of the ocular surface1. An estimated 25 million Americans are reported to have dry eye disease (DED)2, which is a number that will only increase with the U.S. aging population3. The only treatment currently available in the U.S. targets inflammation on the ocular surface. Because dry eye is a complicated disease that encompasses many conditions of the eye, diversified ways to treating the disease are necessary. Some recent studies suggests that some Dry Eye symptoms are caused by corneal cold thermoreceptors (such as TRPM8) chronically firing at below-normal thresholds. It thus logically follows that dry eye patients could be distinguished from normal patients by possessing higher symptom responses secondary to topical application of menthol, a potent agonist of TRPM8. If dry eye patients indeed have lower threshold firing of TRPM8, agonizing TRPM8 with menthol will elicit a more severe symptom response, given equal concentrations across populations.

To fully elucidate this relationship between TRPM8 agonists, sensation, and tear film cooling, two dry eye populations will be tested - one population which has exhibited symptom response to a previous dry eye agent, and one population with no symptom response to the same agent.

ELIGIBILITY:
Inclusion Criteria:

1. Be male or female of any race, at least 18 years of age at Visit 1.
2. Have provided verbal and written informed consent.
3. Have a best corrected visual acuity of +0.70 logMAR or better in both eyes at Visit 1, as assessed by Early Treatment of Diabetic Retinopathy Study (ETDRS) chart.
4. Qualify for exactly one of the three cohorts.

Exclusion Criteria:

1. Have any contraindications to the use of Systane® Ultra, or Rohto® Hyrda, or its components (including Menthol).
2. Have a known allergy to the study medications or their components.
3. Have any clinically significant slit lamp findings at Visit 1, including active blepharitis, meibomian gland dysfunction (MGD), lid margin inflammation or ocular allergies that requires therapeutic treatment and/or, in the opinion of the investigator, may interfere with the study parameters.
4. Be diagnosed with an ongoing ocular infection (bacterial, viral or fungal), or active ocular inflammation (e.g., follicular conjunctivitis) at Visit 1.
5. Have a history of laser in situ keratomileusis (LASIK) surgery in either eye.
6. Have had any ocular surgical procedure within 12 months prior to Visit 1.
7. Have used contact lenses within 30 days prior to Visit 1 and for the duration of the study.
8. Have used any topical ocular prescription (including medications for glaucoma) or over-the-counter (OTC) solutions, artificial tear substitutes, gels or scrubs within 24 hours prior to Visit 1 and for the duration of the study, except for the study drops.
9. Have an uncontrolled systemic disease.
10. Be a woman who is pregnant, nursing an infant, or planning a pregnancy.
11. Have a condition or is in a situation that, in the opinion of the investigator, may put the patient at significant risk, may confound the study results, or may interfere significantly with the patients' participation in the study.
12. Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days prior to Visit 1.
13. Currently have any punctal occlusions in either eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Lane, Study Director — Ora Clinical

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Corcoran P, Hollander DA, Ousler GW 3rd, Angjeli E, Rimmer D, Lane K, Abelson MB. Dynamic Sensitivity of Corneal TRPM8 Receptors to Menthol Instillation in Dry Eye Versus Normal Subjects. J Ocul Pharmacol Ther. 2017 Nov;33(9):686-692. doi: 10.1089/jop.2017.0050. Epub 2017 Sep 21. PMID 28933582

RESULTS

PARTICIPANT FLOW:
Groups:
- Dry Eye Participants: Participants with dry eye received 1 drop of menthol-containing over the counter eye drop (Rohto [r] Hydra) in one eye and 1 drop of comparator treatment (Systane [r] Ultra), which did not contain menthol, in the other.
- Normal Participants: Participants who did not have dry eye received 1 drop of menthol-containing over the counter eye drop (Rohto [r] Hydra) in one eye and 1 drop of comparator treatment (Systane [r] Ultra), which did not contain menthol, in the other.
Period: Overall Study
Arm/Group | Dry Eye Participants | Normal Participants
Started | 33 | 15
Completed | 33 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dry Eye Participants | Normal Participants | Total
Number analyzed (Participants) | 33 | 15 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 15 | 37
  >=65 years | 11 | 0 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (8.6) | 53.5 (7.6) | 58.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 9 | 33
  Male | 9 | 6 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 29 | 14 | 43
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Sum of the Cooling Scale For Rohto (r) Hydra
Description: Participants completed the cooling scale after receiving 1 dose of Rohto (r) Hydra at 6 time points (0, 0.5, 1, 2, 3, and 4 minutes post-treatment), and the scores were summed across these time points. The cooling scale was on a scale of 0 to 10, where 0=not cool and 10=very cool. The summed total was on a scale of 0= not cool and 60=very cool.
Time Frame: 4 Minutes
Population: All Participants Population- all participants who received both study treatments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dry Eye Participants | Normal Participants
Number analyzed (Participants) | 33 | 15
units on a scale | 24.6 (12.2) | 12.1 (9.3)

2. Secondary Outcome: Sum of the Cooling Scale For Systane (r) Ultra
Description: Participants completed the cooling scale after receiving 1 dose of Systane (r) Ultra at 6 time points (0, 0.5, 1, 2, 3, and 4 minutes post-treatment), and the scores were summed across these time points. The cooling scale was on a scale of 0 to 10, where 0=not cool and 10=very cool. The summed total was on a scale of 0= not cool and 60=very cool.
Time Frame: 4 minutes
Population: All Participants Population- all participants who received both study treatments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dry Eye Participants | Normal Participants
Number analyzed (Participants) | 33 | 15
units on a scale | 12.6 (9.4) | 5.2 (6.1)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the signing of the informed consent form to the end of the study, approximately 1 month.
Groups:
- Dry Eye Participants: Participants with dry eye received 1 drop of menthol-containing over the counter eye drop (Rohto [r] Hydra) in one eye and 1 drop of comparator treatment (Systane [r] Ultra), which did not contain menthol.
- Normal Participants: Participants who did not have dry eye received 1 drop of menthol-containing over the counter eye drop (Rohto [r] Hydra) in one eye and 1 drop of comparator treatment (Systane [r] Ultra), which did not contain menthol.
Arm/Group | Dry Eye Participants | Normal Participants
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/15
Other Adverse Events (participants affected / at risk) | 0/33 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No